CLINICAL TRIAL: NCT06524661
Title: Anterior Segment Changes After Pars Plana Vitrectomy With Silicone Oil Tamponade And After Silicone Oil Evacuation Using AS-OCT.
Brief Title: Anterior Segment Changes After Pars Plana Vitrectomy With SO Using AS-OCT
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohab Mohamed Khairy Talaat, Mohab Mohamed Khairy Talaat, Minia University
Other Study IDs: AS-OCT after PPV with SO
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Glaucoma
Keywords: ASOCT; Glaucoma; Silicone; vitrectomy; angle
MeSH Terms: conditions — Glaucoma | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with RRD who underwent pars plana vitrectomy with: AS-oct measuring the anterior chamber angle and corneal changes after pars plana vitrectomy with silicone oil 1000cs injection
  Interventions: Device: AS-OCT after vitrectomy

INTERVENTIONS:
Device: AS-OCT after vitrectomy — AS-OCT is a light based imaging technique of the anterior segment of the eye in this study it is used to measure the anterior chamber angle changes after pars plana vitrectomy.
  Other Names: vitrectomy, silicone oil 1000cs, silicone oil evacuation

SUMMARY:
To evaluate changes in ACA induced by pars plana vitrectomy with SO 1000cs injection in vitreo-retinal surgery in phakic eyes using AS-OCT and changes in the IOP preoperatively, post-operatively and post-silicone oil evacuation.

DETAILED DESCRIPTION:
Abstract Introduction Ocular hypertension and secondary glaucoma are relatively common and serious complications in silicone filled eyes which may end in blindness. Reports have described the percentage of incidence to be within 3 - 30 % of silicon filled eye which are complicated with secondary glaucoma. [1] Aim of study Evaluation of changes in anterior chamber angle and intra-ocular pressure (IOP) in patients with rhegmatogenous retinal detachment (RRD) who underwent pars plana vitrectomy (PPV) with silicone oil (SO) 1000cs tamponade and after silicone oil evacuation.

Population The study was a prospective interventional study. The study included 30 eyes from 30 patients with rhegmatogenous retinal detachment (RRD) who are going to undergo PPV with SO injection. The study was conducted at Ophthalmology department, Minia University Hospital in Egypt between April 2023 and April 2024.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with rhegmatogenous retinal detachment who are going to undergo vitreoretinal surgery with silicone oil 1000cs injection as tamponade

Exclusion Criteria:

* Patients with history of intraocular surgery, laser therapy or intravitreal injection.
* Patients with significant corneal opacity.
* Patients with ocular diseases as retinal vein occlusion, uveitis and proliferative diabetic retinopathy.
* Patients with preexisting glaucoma or family history of glaucoma.
* Patients with nystagmus.
* Patient with tractional retinal detachment, exudative retinal detachment or intraocular foreign body.
* Patients with anterior chamber abnormalities including posterior synechia, peripheral anterior synechia, hyphaema and iris abnormalities.
* Patients with severe proliferative vitreoretinopathy grade C or more.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are phakic with rhegmatogenous retinal detachment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Assessement of the changes in anterior chamber angle after vitrectomy with silicone oil injection | postoperative evaluation for 3 months duration (5 visits pre-ppv then one week, one month, three months )
  Evaluation of changes in the anterior chamber angle parameters after vitrectomy with silicone oil 1000cs injection.
  The measures include AOD 500, TISA 500, ACA and CCT The measuring tool is AS-OCT (anterior segment optical coherent topography)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine ,Minia university, Minya, Egypt

REFERENCES:
- [Background] Calik B, Ozturk M, Serdarogullari H, Elcioglu M. Evaluation of anterior segment parameters using pentacam in silicone oil-injected patients after pars plana vitrectomy. Indian J Ophthalmol. 2013 Nov;61(11):621-5. doi: 10.4103/0301-4738.123137. PMID 24343592